CLINICAL TRIAL: NCT01548482
Title: A Phase I Trial of AMG 386 and Temsirolimus in Advanced Solid Tumors With an Expansion Cohort in Uterine Cancer, Renal Cell Carcinoma and Carcinoid Tumor
Brief Title: Trebananib And Temsirolimus in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02848; NCI-2012-02848 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000728823; PJC-008 (Other: University Health Network-Princess Margaret Hospital); 9041 (Other: CTEP); U01CA132123 (NIH); UM1CA186644 (NIH)
Record Dates: First submitted 2012-02-24; First posted 2012-03-08 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-05

CONDITIONS: Adult Solid Neoplasm; Lung Carcinoid Tumor; Recurrent Digestive System Neuroendocrine Tumor G1; Recurrent Renal Cell Carcinoma; Recurrent Uterine Corpus Sarcoma; Stage III Renal Cell Cancer; Stage IIIB Uterine Sarcoma; Stage IIIC Uterine Sarcoma; Stage IV Renal Cell Cancer; Stage IVA Uterine Sarcoma; Stage IVB Uterine Sarcoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — temsirolimus; Sirolimus; trebananib

ARMS (1):
- Treatment (trebananib, temsirolimus) (Experimental): Patients receive trebananib IV over 60 minutes and temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus; Biological: Trebananib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
Biological: Trebananib — Given IV
  Other Names: AMG 386; Angiopoietin 1/2-Neutralizing Peptibody AMG 386

SUMMARY:
This phase I trial studies the side effects and the best dose of trebananib and temsirolimus when given together in treating patients with solid tumors that are metastatic or cannot be removed by surgery. Trebananib may stop the growth of tumor cells by blocking blood flow to the tumor. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving trebananib with temsirolimus may be an effective treatment for solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RP2D) and safety profile of AMG 386 (trebananib) in combination with temsirolimus in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To evaluate pharmacodynamic (PD) effects of both drugs when administered in combination, with the goal of identifying potential predictive and PD markers that need further exploration and validation in future trials.

II. To explore preliminary anti-tumor activity of both drugs when administered at the RP2D to patients with advanced endometrial cancer, renal cell carcinoma, or carcinoid tumor.

OUTLINE: This is a dose-escalation study of trebananib.

Patients receive trebananib intravenously (IV) over 60 minutes and temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* DOSE ESCALATION COHORTS: Patients must have histologically or cytologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* DOSE EXPANSION COHORTS: Patients must have histologically and/or cytologically confirmed uterine cancer, renal cell cancer or carcinoid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* DOSE ESCALATION COHORTS: No limitation on prior therapy; however, there must be at least a 4 week interval between initiation of study treatment and any prior radiotherapy or systemic therapy, 6 weeks if the last regimen included carmustine (BCNU) or mitomycin C; exceptions may be made however, for low dose, non-myelosuppressive radiotherapy for symptomatic palliation; please contact the study coordinator at the Princess Margaret Hospital (PMH) Phase I Consortium Central Office or the principal investigator if any questions arise about interpretation of this criterion
* EXPANSION COHORTS:

  * Uterine cancer: Patients diagnosed with uterine cancer will be eligible provided they have received at least one prior line of chemotherapy for recurrent or metastatic disease unless the investigator feels that cytotoxic chemotherapy is contraindicated; prior hormonal treatment will be allowed; prior anti-angiogenic agents and prior treatment with agents targeting phosphatidylinositol 3-kinase (PI3K)- protein kinase B (AkT)- mammalian target of rapamycin (mTOR) pathway are not allowed
  * Renal cell cancer: Patients diagnosed with renal cell cancer (RCC) will be required to have received at least one prior line anti- vascular endothelial growth factor (VEGF)/ receptor (R) treatment (i.e. bevacizumab, sunitinib, and/or sorafenib); prior treatment with agents targeting PI3K-Akt-mTOR pathway is not allowed
  * Carcinoid tumor: Patients diagnosed with carcinoid tumor must have demonstrated radiographic evidence of disease progression within six months prior to enrollment; prior and/or concurrent long-acting somatostatin analogue therapy is allowed; if patient is continued on a long-acting somatostatin analogue, a stable dose for >= 2 months prior to study entry is required with documentation of progressive disease on current dose; prior radiolabeled octreotide therapy is allowed; prior regional treatments for liver metastasis are permitted including:

    * Selective internal radiation therapy (i.e. brachytherapy, radiolabeled microsphere embolization, etc)
    * Hepatic artery chemoembolization
    * Hepatic artery embolization
    * Hepatic artery infusional chemotherapy
    * Radiofrequency ablation
  * Patients must be > 12 weeks from regional treatments and show progressive disease in the liver after regional therapy or must have measurable disease outside the liver; patients may have received one prior line of anti-VEGF/R treatment (e.g. bevacizumab, sunitinib, and/or sorafenib); prior treatment with agents targeting PI3K-Akt-mTOR pathway is not allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3.0 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 90 g/L (or >= 9 g/dL)
* Total bilirubin =< institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal if no known liver metastasis or =< 5 x institutional upper limit of normal if known liver metastasis
* Partial thromboplastin time (PTT) or activated PTT (aPTT) =< 1.5 x ULN per institutional laboratory range and international normalized ratio (INR) =< 1.5
* Creatinine =< institutional ULN OR creatinine clearance > 40 mL/min per 24 hours (h) urine collection or calculated according to the Cockcroft-Gault formula
* Urinary protein =< 30 mg/dL in urinalysis or =< 1 + on dipstick, unless quantitative protein is < 1000 mg in a 24 h urine sample
* Total cholesterol < 400 mg/dL (or < 10.34 mmol/L)
* Serum triglyceride level < 500 mg/dL (or < 5.7 mmol/L)
* Generally well-controlled blood pressure with systolic blood pressure =< 140 mm Hg AND diastolic blood pressure =< 90 mm Hg prior to enrollment; the use of anti-hypertensive medications to control hypertension is permitted
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and 6 months after completion of AMG386 and/or temsirolimus administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of AMG386 and/or temsirolimus administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of central nervous system metastases
* History of venous or arterial thromboembolism within 12 months prior to enrollment/randomization; patients requiring ongoing anticoagulation with therapeutic dosages of low molecular weight heparin or warfarin are excluded
* History of clinically significant bleeding within 6 months of enrollment/randomization
* Unresolved toxicities from prior systemic therapy that are Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 >= grade 2 in severity except alopecia
* Currently or previously treated with AMG 386, or other molecules that inhibit the angiopoietins or TEK tyrosine kinase, endothelial (Tie2) receptor
* Clinically significant cardiovascular disease within 12 months prior to enrollment/randomization, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication or placement of percutaneous transluminal coronary angioplasty/stent
* Major surgery within 28 days prior to enrollment or still recovering from prior surgery
* Minor surgical procedures, except placement of tunneled central venous access device within 3 days (7 days if with VEGF inhibitor) prior to randomization/enrollment
* Treatment within 30 days prior to enrollment with strong immune modulators, including but not limited to systemic cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, methotrexate, azathioprine, rapamycin, thalidomide, lenalidomide, and targeted immune modulators such as abatacept (CTLA-4-Ig), adalimumab, alefacept, anakinra, belatacept (LEA29Y), efalizumab, etanercept, infliximab, or rituximab
* Non-healing wound, ulcer (including gastrointestinal), or fracture
* Subject not consenting to the use of highly effective contraceptive precautions (e.g., double barrier method [i.e., condom plus diaphragm]) during the course of the study and for 6 months after administration of the last study medication
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AMG 386 or temsirolimus
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have not yet completed at least 21 days (30 days for prior monoclonal antibody therapy) since ending other investigational device or drug trials, or who are currently receiving other investigational treatments
* Temsirolimus is a cytochrome P450 3A4 (CYP3A4) substrate; patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with AMG 386; these potential risks may also apply to temsirolimus
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients with pre-existing clinically significant pulmonary infiltrates of unknown origin
* Patients with an indwelling peritoneal or pleural catheter that is used to manage malignant effusions
* Known intra-abdominal inflammatory process or serious gastrointestinal ulceration
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No gastric or esophageal varices
* Patients with primary bowel tumors in situ or recurrent disease at bowel anastomosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
RP2D of trebananib and temsirolimus defined as the dose level at which =< 1/6 patients experienced dose-limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) CTCAE version 4.0 | 28 days
Safety profile of trebananib and temsirolimus as assessed by NCI CTCAE version 4.0 | Up to 30 days
  Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. Adverse events will be summarized using all adverse events experienced, although a subanalysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to one or both study treatments.

SECONDARY OUTCOMES:
Objective response to treatment assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 | Up to 30 days
  Predictors of clinical outcomes will be investigated using logistic regression, Cox proportional hazards regression and/or generalized estimating equations as appropriate.
PD effects of both drugs when administered in combination | Course 1 days 1, 3, and 8 and course 2 day 1
  Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (3):
- Canada (3):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario